CLINICAL TRIAL: NCT02742467
Title: Comparison of Three Combination Therapies in Lowering Blood Pressure in Black Africans
Acronym: Creole
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Abuja (Other)
Collaborators: Imperial College London (Other); University of Cape Town (Other); Hôpital Edouard Herriot (Other); University of Nairobi (Other); University College Hospital, Ibadan (Other); Hospital General De Douala (Other); Mulago Hospital, Uganda (Other)
Responsible Party: Principal Investigator, Dr. Dike Ojji, Dr, University of Abuja
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Project8264
Record Dates: First submitted 2016-04-14; First posted 2016-04-19 (Estimated); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Perindopril; Amlodipine; Hydrochlorothiazide

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1 (Experimental): Perindopril plus Amlodipine at a dose of 4mg/5mg once daily for two months and 8mg/10mg once daily for the remaining four months.
  Interventions: Drug: Perindopril plus Hydrochlorothiazide; Drug: Amlodipine plus Hydrochlorothiazide
- 2 (Active Comparator): Perindopril Plus Hydrochlorothiazide at a dose of 4mg/12.5mg and 8mg/25mg once daily for the remaining four months.
  Interventions: Drug: Perindopril plus Amlodipine; Drug: Amlodipine plus Hydrochlorothiazide
- 3 (Active Comparator): Amlodipine plus Hydrochlorothiazide 5mg/12.5mg for two months and 10mg/25mg for the remaining four months.
  Interventions: Drug: Perindopril plus Amlodipine; Drug: Perindopril plus Hydrochlorothiazide

INTERVENTIONS:
Drug: Perindopril plus Amlodipine — Group 1
  Arms: 2; 3
Drug: Perindopril plus Hydrochlorothiazide — Group 2
  Arms: 1; 3
Drug: Amlodipine plus Hydrochlorothiazide — Group 3
  Arms: 1; 2

SUMMARY:
The creole study is a A Multi-centre, multinational, randomised single-blind, parallel group, three-armed superiority trial which is aimed at comparing the efficacy of three "free" combinations of two anti-hypertensive agents on 24 hour ambulatory systolic blood pressure (ASBP) in black African hypertensive patients.

DETAILED DESCRIPTION:
The CREOLE trial will be performed at ten investigational sites in six countries in Sub-Saharan Africa which include Cameroun, Kenya, Mozambique, Nigeria, South Africa and Uganda. Subjects will be randomised to one of three treatments which are Perindopril plus Amlodipine or Perindopril plus Hydrochlorothiazide or Amlodipine plus Hydrochlorothiazide.Patients will commence treatment at a starting dose of Amlodipine plus Hydrochlorothiazide 5/12.5 mg or Amlodipine plus Perindopril 5/4 mg or Perindopril/Hydrochlorothiazide 4/12.5 mg. These doses will increase at the two months visit, to Amlodipine/Hydrochlorothiazide 10/25 mg or AmlodipinePperindopril 10/8mg or Perindopril/Hydrochlorothiazide 8/25 mg.

The patients will have ambulatory blood pressure monitoring at randomization and at six months and office blood pressure measurements at randomization and at two-month, 4-month and six-month visits.The overall aim is to discover the best combination of front-line anti-hypertensive medications for black patients residing in sub-Saharan Africa.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Sitting SBP ≥140 mm Hg and < 160 mmHg on one antihypertensive agen or
* Sitting SBP ≥ 150 mm Hg and < 180 mm Hg on no antihypertensive treatment.

Exclusion Criteria:

* Congestive heart failure (clinically defined).
* Serum creatinine levels greater than 170 µmol/l or estimated glomerular filtration rate (eGFR) < 30 ml/min.
* History of coronary heart disease (i.e., chronic stable angina, myocardial infarction or acute coronary syndrome).
* History of a stroke or other cerebrovascular accident (i.e. transient ischaemic attack or reversible ischaemic neurological deficit).
* Known or suspected secondary hypertension.
* Any other concomitant illness, physical or mental impairment that could interfere with the effective conduct of the study.
* Pregnancy or those of child-bearing age who are not taking reliable contraception.
* Patients with a history of intolerance to any of the study medications for example angioedema or dry cough with angiotensin converting enzyme inhibitors.
* Patients on maximum dose of any of the study medications as monotherapy (i.e. amlodipine 10 mg/day or hydrochlorothiazide 25 mg/day or perindopril 8 mg/day)
* Gout.
* Serum potassium < 3.5mmol/L at screening.

Ages: 30 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 702 (Actual)
Dates: Start 2017-06-07 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Ambulatory blood pressure | six months
  Change in ambulatory systolic blood pressure measurement from baseline to 6 months from will be determined.

SECONDARY OUTCOMES:
Assessment of ambulatory diastolic blood pressure | six months
  Change in 24 hour ambulatory diastolic blood pressure between randomisation and 6 months
Clinic systolic and diastolic blood pressure | Six months
  Change in clinic systolic and diastolic blood pressure will be difference in values between randomisation and 6 months
Night time and day time blood pressure | Six months
  Change in daytime and night time blood pressure
Blood pressure control | Six months
  change in BP variability measured will be measured by ambulatory blood pressure
Blood pressure control | Two months and six months
  Proportion of patients who achieve BP control (defined as clinic BP < 140/90 mmHg) after 6 months
Response to study medications | Two months and six months
  Proportion of "responders" (defined as clinic BP reduction > 20mmHg SBP and >10 mmHg DBP) from randomisation to 6 months
Change in values of micro- and macro-albuminuria | Six months
  Change in micro- and macro-albuminuria will be measured from randomisation to 6 months
Fasting blood sugar variation | Six months
  Change in fasting blood sugar which will be from randomisation to 6 months
Fasting lipid profile variation | Six months
  Change in fasting lipid profile between from randomisation to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Neil Poulter, MD, MSc, Study Director — Imperial College London; Bongani Mayosi, DPhil, Study Chair — University of Cape Town
Locations (1):
- University of Abuja Teaching Hospital, Abuja, Federal Capital Territory, Nigeria

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Ingabire PM, Ojji DB, Rayner B, Ogola E, Damasceno A, Jones E, Dzudie A, Ogah OS, Poulter N, Sani MU, Barasa FA, Shedul G, Mukisa J, Mukunya D, Wandera B, Batte C, Kayima J, Pandie S, Mondo CK; CREOLE Study Investigators. High prevalence of non-dipping patterns among Black Africans with uncontrolled hypertension: a secondary analysis of the CREOLE trial. BMC Cardiovasc Disord. 2021 May 22;21(1):254. doi: 10.1186/s12872-021-02074-7. PMID 34022790
- [Derived] Ojji DB, Mayosi B, Francis V, Badri M, Cornelius V, Smythe W, Kramer N, Barasa F, Damasceno A, Dzudie A, Jones E, Mondo C, Ogah O, Ogola E, Sani MU, Shedul GL, Shedul G, Rayner B, Okpechi IG, Sliwa K, Poulter N; CREOLE Study Investigators. Comparison of Dual Therapies for Lowering Blood Pressure in Black Africans. N Engl J Med. 2019 Jun 20;380(25):2429-2439. doi: 10.1056/NEJMoa1901113. Epub 2019 Mar 18. PMID 30883050